CLINICAL TRIAL: NCT03630705
Title: Safety and Immunogenicity of a 3-Dose Schedule of an Investigational Quadrivalent Meningococcal Conjugate Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers
Brief Title: Safety and Immunogenicity of a Quadrivalent Meningococcal Conjugate Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers in the Russian Federation and Mexico
Acronym: MET33
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MET33; U1111-1183-6409 (Registry Identifier: ICTRP)
Record Dates: First submitted 2018-08-03; First posted 2018-08-15 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers (Meningococcal Infection)
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines; Measles-Mumps-Rubella Vaccine; 13-valent pneumococcal vaccine; Tetanus Toxoid; Elements; Vaccines; Pentavac; Hepatitis B Vaccines; Engerix-B; Rotavirus Vaccines; RotaTeq; DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: MenACYW Conjugate Vaccine (Mexico) (Experimental): Participants aged 2 months (at the time of enrollment) received Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus toxoid (MenACYW) Conjugate vaccine at the age of Months 2, 6, and 12 along with Prevnar 13®, Hexacima®, vaccines at the age of Months 2, 4, 6 and 12; RotaTeq® vaccine at the age of Months 2, 4 and 6 and measles, mumps, rubella (MMR®II) vaccine at the age of Month 12.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Rotavirus Vaccine, Live, Pentavalent; Biological: Diphtheria, tetanus, pertussis (acellular component), hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b conjugate vaccine
- Group 2: Menveo® (Mexico) (Active Comparator): Participants aged 2 months (at the time of enrollment) received Menveo® vaccine at the age of Months 2, 4, 6, and 12 along with Prevnar 13®, Hexacima® vaccines at the age of Months 2, 4, 6 and 12; RotaTeq® vaccine at the age of Months 2, 4 and 6, and MMR®II vaccine at the age of Month 12.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Rotavirus Vaccine, Live, Pentavalent; Biological: Diphtheria, tetanus, pertussis (acellular component), hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b conjugate vaccine
- Group 3: MenACYW Conjugate Vaccine (Russian Federation) (Experimental): Participants aged 2 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of Months 3, 6, and 12 along with Prevnar 13® vaccine at the age of Months 2, and 4.5; Pentaxim® vaccine at the age of Months 3, 4.5, and 6; ENGERIX-B® vaccine at the age of Month 6 and MMR vaccine at the age of Month 12.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Diphtheria, Tetanus, Pertussis (Acellular, Component) Poliomyelitis (inactivated) Vaccine, and Haemophilus influenza type b Conjugate Vaccine; Biological: Hepatitis B Vaccine
- Group 4: Routine Pediatric Vaccines (Russian Federation) (Other): Participants aged 2 months (at the time of enrollment) received Prevnar 13® vaccine at the age of Months 2, and 4.5; Pentaxim® vaccine at the age of Months 3, 4.5, and 6; ENGERIX-B® vaccine at the age of Month 6 and MMR vaccine at the age of Month 12.
  Interventions: Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Diphtheria, Tetanus, Pertussis (Acellular, Component) Poliomyelitis (inactivated) Vaccine, and Haemophilus influenza type b Conjugate Vaccine; Biological: Hepatitis B Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — Pharmaceutical form: Liquid solution Route of administration : Intramuscular
  Arms: Group 1: MenACYW Conjugate Vaccine (Mexico); Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Biological: Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine — Pharmaceutical form: Lyophilized powder combined with liquid component Route of administration : Intramuscular
  Other Names: Menveo®
  Arms: Group 2: Menveo® (Mexico)
Biological: Measles, Mumps, and Rubella Virus Vaccine Live — Pharmaceutical form: Lyophilized live virus vaccine Route of administration : Subcutaneous
  Other Names: M-M-R®II
Biological: Pneumococcal 13-valent Conjugate Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Other Names: Prevnar 13®
Biological: Diphtheria, Tetanus, Pertussis (Acellular, Component) Poliomyelitis (inactivated) Vaccine, and Haemophilus influenza type b Conjugate Vaccine — Pharmaceutical form: Powder and suspension for injection Route of administration: Intramuscular
  Other Names: Pentaxim®
  Arms: Group 3: MenACYW Conjugate Vaccine (Russian Federation); Group 4: Routine Pediatric Vaccines (Russian Federation)
Biological: Hepatitis B Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Other Names: ENGERIX-B®
  Arms: Group 3: MenACYW Conjugate Vaccine (Russian Federation); Group 4: Routine Pediatric Vaccines (Russian Federation)
Biological: Rotavirus Vaccine, Live, Pentavalent — Pharmaceutical form: Oral solution Route of administration: Oral
  Other Names: RotaTeq®
  Arms: Group 1: MenACYW Conjugate Vaccine (Mexico); Group 2: Menveo® (Mexico)
Biological: Diphtheria, tetanus, pertussis (acellular component), hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b conjugate vaccine — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Other Names: Hexacima®
  Arms: Group 1: MenACYW Conjugate Vaccine (Mexico); Group 2: Menveo® (Mexico)

SUMMARY:
Primary Objective:

1. To describe the vaccine seroprotection (antibody titer greater than or equal to [>=] 1:8) to the antigens (meningococcal serogroups A, C, Y, and W) present in MenACYW Conjugate vaccine or Menveo® measured by serum bactericidal assay using human complement (hSBA), for Groups 1 and 2 when administered concomitantly with routine pediatric vaccines in healthy infants and toddlers in Mexico.
2. To describe the vaccine seroprotection (antibody titer >=1:8) to the antigens (meningococcal serogroups A, C, Y, and W) present in MenACYW Conjugate vaccine measured by hSBA, for Group 3, when administered concomitantly with routine pediatric vaccines in healthy infants and toddlers in the Russian Federation.

Secondary Objective:

1. To describe hSBA vaccine seroresponse to the antigens (meningococcal serogroups A, C, Y, and W) 30 days after the last vaccination of the infant series, when administered concomitantly with routine pediatric vaccines in healthy infants and toddlers in Mexico and Russian Federation (RF).
2. To describe immunogenicity profile of routine pediatric vaccines when administered concomitantly with MenACYW Conjugate vaccine or Menveo®; or when administered alone.
3. To describe hSBA antibody responses against meningococcal serogroups A, C, Y, and W when MenACYW Conjugate vaccine and Menveo® are administered concomitantly with routine pediatric vaccines in Mexico and RF.
4. To describe antibody titers to the antigens present in MenACYW Conjugate vaccine and Menveo®, before the first vaccination and 30 days after the last vaccination of the infant series and in the second year of life, when administered concomitantly with routine pediatric vaccines in a subset of participants in Mexico and RF.

DETAILED DESCRIPTION:
Study duration per participant was approximately 12 months.

ELIGIBILITY:
Inclusion criteria:

An individual must fulfill all of the following criteria in order to be eligible for trial enrollment:

* Infants 2 months of age (60 to 89 days of age) on the day of the first study visit.*
* Born after a full-term pregnancy, with an estimated gestation age >= 37 weeks and a birth weight >= 2.5 kilograms.
* Informed consent form has been signed and dated by the parent(s) or guardian(s), as required by local regulations.†
* Participant and parent/guardian were able to attend all scheduled visits and to comply with all trial procedures.
* In good health as determined by medical history and physical assessment.
* For the Russian Federation: The participant's parents were able to verbally report or provide written documentation that the participant's mother was hepatitis B antigen negative during pregnancy with the participant.

  * * "2 months" means from the 2nd month after birth to the day before the 3rd month after birth (2 months to 2 months 29 days); "60 days" means from the 60th day after birth to the day before the 90th day after birth (60 to 89 days).

    * † In the Russian Federation, as per local regulations, only the participant's parent(s) were entitled to sign an informed consent form. A child under the responsibility of a guardian would not be included in the study.

Exclusion criteria:

An individual fulfilling any of the following criteria was to be excluded from trial enrollment:

* Participation at the time of study enrollment or in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks before and/or following any trial vaccination except for influenza vaccination, which may be received at a gap of at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., meningitis polysaccharide or meningitis Conjugate vaccine containing serogroups A, C, Y, or W; or meningococcal B serogroup-containing vaccine).
* Previous vaccination against diphtheria, tetanus, pertussis, Haemophilus influenzae type b (Hib), poliovirus, rotavirus, Streptococcus pneumoniae, measles, mumps, rubella, and / or varicella.
* For Mexico: More than 1 previous dose of hepatitis B vaccine.
* Receipt of immune globulins, blood or blood-derived products since birth.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) since birth.
* Family history of congenital or hereditary immunodeficiency until the immune competence of the potential vaccine recipient is demonstrated.
* Individuals with blood dyscrasias, leukemia, lymphoma of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Individuals with active tuberculosis.
* History of any Neisseria meningitidis infection, confirmed either clinically, serologically, or microbiologically.
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, hepatitis A, measles, mumps, rubella, Haemophilus influenzae type b, Streptococcus pneumoniae, and /or rotavirus infection / disease.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease).
* History of intussusception.
* History of any neurologic disorders, including seizures (febrile and non-febrile) and progressive neurologic disorders.
* History of Guillain-Barré syndrome.
* Known systemic hypersensitivity to any of the vaccine components or to latex, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances, including neomycin, gelatin, and yeast.
* Verbal report of thrombocytopenia contraindicating intramuscular vaccination in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion.
* Receipt of oral or injectable antibiotic therapy within 72 hours of the first blood draw.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0 degree Celsius [°C]). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

  * For the Russian Federation, febrile illness was defined as temperature >= 37°C. A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 525 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Mexico (3):
  - Investigational Site Number :4840001, Acapulco de Juárez, Guerrero
  - Investigational Site Number :4840002, Mexico City, Mexico City
  - Investigational Site Number :4840003, Tlaltizapán, Morelos
- Russia (8):
  - Investigational Site Number :6431018, Gatchina, Leningradskaya Oblast'
  - Investigational Site Number :6431008, Krasnodar
  - Investigational Site Number :6431004, Perm
  - Investigational Site Number :6431007, Saint Petersburg
  - Investigational Site Number :6431010, Saint Petersburg
  - Investigational Site Number :6431001, Saint Petersburg
  - Investigational Site Number :6431006, Samara
  - Investigational Site Number :6431002, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted from 17 October 2018 to 18 February 2022 at 11 active sites in Mexico and the Russian Federation.
Pre-assignment Details: A total of 525 participants were enrolled and randomized in the study.
Groups:
- Group 2: Menveo® Vaccine (Mexico): Participants aged 2 months (at the time of enrollment) received Menveo® vaccine at the age of Months 2, 4, 6, and 12 along with Prevnar 13®, Hexacima® vaccines at the age of Months 2, 4, 6 and 12; RotaTeq® vaccine at the age of Months 2, 4 and 6, and MMR®II vaccine at the age of Month 12.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Started | 200 | 100 | 150 | 75
Vaccinated at the Age of 2 Months | 200 | 100 | 150 | 75
Vaccinated at the Age of 3 Months (Group 1 and 2 participants did not receive any vaccination at the age of 3 months.) | 0 | 0 | 149 | 75
Vaccinated at the Age of 4 Months (Group 3 and 4 participants did not receive any vaccination at the age of 4 months.) | 195 | 96 | 0 | 0
Vaccinated at the Age of 4.5 Months (Group 1 and 2 participants did not receive any vaccination at the age of 4.5 months.) | 0 | 0 | 149 | 75
Vaccinated at the Age of 6 Months | 194 | 95 | 149 | 75
Vaccinated at the Age of 12 Months | 192 | 92 | 148 | 75
Safety Analysis Set (Safety analysis set (SafAS) included those participants who had received at least 1 dose of the study vaccine and had any safety data available. All participants had their safety analyzed after each dose according to the vaccine they actually received at that dose.) | 201 (One participant of arm 'Group 2: Menveo® (Mexico)' received MenACYW Conjugate vaccine at the age of 2 months and thus included in the safety analysis of arm 'Group 1: MenACYW Conjugate Vaccine (Mexico)'.) | 99 | 150 | 75
Completed | 190 | 92 | 148 | 75
Not Completed | 10 | 8 | 2 | 0
Not completed — Withdrawal by Parent/Guardian | 9 | 6 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine (Mexico): Participants aged 2 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of Months 2, 6, and 12 along with Prevnar 13®, Hexacima®, vaccines at the age of Months 2, 4, 6 and 12; RotaTeq® vaccine at the age of Months 2, 4 and 6 and MMR®II vaccine at the age of Month 12.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation) | Total
Number analyzed (Participants) | 200 | 100 | 150 | 75 | 525
Age, Continuous [Mean (Standard Deviation); unit: months] | 2.2 (0.24) | 2.3 (0.25) | 2.4 (0.28) | 2.4 (0.29) | 2.3 (0.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 54 | 69 | 48 | 271
  Male | 100 | 46 | 81 | 27 | 254
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 166 | 78 | 0 | 0 | 244
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 150 | 75 | 225
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 34 | 22 | 0 | 0 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers Greater Than or Equal to (>=) 1:8 Against Meningococcal Serogroups A, C, Y, and W Following Last Vaccination With MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by serum bactericidal assay using human complement (hSBA) assay. Group 3 data were presented separately.
Time Frame: 30 days after the last vaccination at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on Per-Protocol Analysis Set 2 (PPAS2) defined for accessing ACYW immune response data for participants who received at least 1 dose of study vaccine and had valid post-vaccination serology result of 2nd year of life, with no major protocol violations. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 126 | 60
percentage of participants
  Serogroup A | 97.6 [93.2 to 99.5] | 95.0 [86.1 to 99.0]
  Serogroup C | 99.2 [95.7 to 100] | 93.3 [83.8 to 98.2]
  Serogroup Y: number analyzed (Participants) | 125 | 60
  Serogroup Y | 100 [97.1 to 100] | 100 [94.0 to 100]
  Serogroup W: number analyzed (Participants) | 125 | 60
  Serogroup W | 100 [97.1 to 100] | 100 [94.0 to 100]

2. Primary Outcome: Percentage of Participants With Antibody Titers >=1:8 Against Meningococcal Serogroups A, C, Y, and W Following Last Vaccination With MenACYW Conjugate Vaccine: Group 3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay.
Time Frame: 30 days after the last vaccination at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 96
percentage of participants
  Serogroup A | 89.6 [81.7 to 94.9]
  Serogroup C | 82.3 [73.2 to 89.3]
  Serogroup Y | 80.2 [70.8 to 87.6]
  Serogroup W | 80.2 [70.8 to 87.6]

3. Secondary Outcome: Percentage of Participants Achieving Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W Following Last Vaccination With MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2 (up to the Infant Age of 6 Months)
Description: The hSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination hSBA titers greater than or equal to (>=) 1:16 for participants with pre-vaccination hSBA titers less than (<) 1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >=1:8. Group 3 data were presented separately. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the last vaccination at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on Per-Protocol Analysis Set 1 (PPAS1) defined for accessing ACYW immune response data for participants who received at least 1 dose of study vaccine and had valid post-vaccination serology result of infancy (6 months of age) vaccination stage, with no major protocol deviations. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 176 | 81
percentage of participants
  Serogroup A | 84.7 [78.5 to 89.6] | 58.0 [46.5 to 68.9]
  Serogroup C | 100 [97.9 to 100] | 86.4 [77.0 to 93.0]
  Serogroup Y | 99.4 [96.9 to 100] | 92.6 [84.6 to 97.2]
  Serogroup W | 98.3 [95.1 to 99.6] | 97.5 [91.4 to 99.7]

4. Secondary Outcome: Percentage of Participants Achieving Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W Following Last Vaccination With MenACYW Conjugate Vaccine: Group 3 (up to the Infant Age of 6 Months)
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. The hSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >=1:16 for participants with pre-vaccination hSBA titers <1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >=1:8. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the last vaccination at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 97
percentage of participants
  Serogroup A | 70.1 [60.0 to 79.0]
  Serogroup C | 94.8 [88.4 to 98.3]
  Serogroup Y | 87.6 [79.4 to 93.4]
  Serogroup W | 93.8 [87.0 to 97.7]

5. Secondary Outcome: Geometric Mean Concentration of Pertussis Toxoid (PT) and Filamentous Hemagglutinin (FHA) Antibodies Before Vaccination With Hexacima® Vaccine Administered Along With MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2 (up to the Infant Age of 6 Months)
Description: Geometric mean concentration (GMCs) for PT and FHA were measured by electrochemiluminescent (ECL) assay. Concentration was expressed in terms of titers (1/dilution). Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: Day 0 (before the first vaccination with Hexacima® vaccine) of the infant series (i.e., at the age of 2 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Groups 3 and 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 126 | 60
titers
  PT | 5.36 [4.27 to 6.73] | 8.34 [6.13 to 11.4]
  FHA | 22.0 [17.2 to 28.1] | 39.9 [27.8 to 57.2]

6. Secondary Outcome: Geometric Mean Concentrations of Anti-rotavirus Serum Immunoglobulin A (IgA) Antibodies Before and After RotaTeq® Vaccine Administered Alone or Along With the MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2 (up to the Infant Age of 6 Months)
Description: GMCs of Anti-rotavirus serum IgA antibodies were assessed using enzyme-linked immunosorbent assay (ELISA). Concentrations were measured in terms of units/milliliter (U/mL). Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: Day 0 (before the first vaccination with RotaTeq® vaccine at the age of 2 months) and 30 days after the vaccination with RotaTeq® vaccine at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Groups 3 and 4.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 176 | 81
U/mL
  Day 0 (at the age of 2 months) | 4.24 [3.84 to 4.67] | 4.91 [4.00 to 6.01]
  At the age of 7 months | 621 [496 to 776] | 572 [402 to 815]

7. Secondary Outcome: Geometric Mean Concentration of Anti-pneumococcal Antibodies After Prevnar 13® Vaccine Administered Alone or Along With the MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2 (up to the Infant Age of 6 Months)
Description: GMCs of anti-pneumococcal antibodies was assessed by electrochemiluminscent (ECL) assay. GMCs of Prevnar 13 serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F were reported. Concentration was expressed in terms of titers (1/dilution). Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the vaccination with Prevnar 13® vaccine at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Here, 'Number analyzed'=participants with available data for the specified categories. Data for this outcome measure was not planned to be collected and analyzed for Groups 3 and 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 176 | 81
titers
  Serotype 1: number analyzed (Participants) | 175 | 81
  Serotype 1 | 3.28 [2.95 to 3.64] | 2.75 [2.34 to 3.24]
  Serotype 3: number analyzed (Participants) | 175 | 81
  Serotype 3 | 0.607 [0.553 to 0.665] | 0.498 [0.436 to 0.569]
  Serotype 4: number analyzed (Participants) | 175 | 81
  Serotype 4 | 1.90 [1.73 to 2.08] | 1.63 [1.42 to 1.86]
  Serotype 5: number analyzed (Participants) | 175 | 81
  Serotype 5 | 2.26 [2.04 to 2.52] | 1.91 [1.65 to 2.21]
  Serotype 6A: number analyzed (Participants) | 175 | 81
  Serotype 6A | 4.57 [4.13 to 5.05] | 3.76 [3.30 to 4.29]
  Serotype 6B: number analyzed (Participants) | 175 | 81
  Serotype 6B | 2.64 [2.30 to 3.03] | 1.96 [1.63 to 2.34]
  Serotype 7F: number analyzed (Participants) | 175 | 81
  Serotype 7F | 3.97 [3.64 to 4.33] | 3.62 [3.21 to 4.08]
  Serotype 9V: number analyzed (Participants) | 175 | 81
  Serotype 9V | 2.33 [2.11 to 2.57] | 1.99 [1.72 to 2.31]
  Serotype 14: number analyzed (Participants) | 174 | 81
  Serotype 14 | 9.36 [8.47 to 10.3] | 9.72 [8.18 to 11.5]
  Serotype 18C: number analyzed (Participants) | 175 | 81
  Serotype 18C | 2.24 [2.06 to 2.45] | 1.71 [1.49 to 1.97]
  Serotype 19A: number analyzed (Participants) | 175 | 81
  Serotype 19A | 2.45 [2.19 to 2.74] | 1.95 [1.72 to 2.21]
  Serotype 19F: number analyzed (Participants) | 175 | 81
  Serotype 19F | 3.55 [3.20 to 3.94] | 2.83 [2.42 to 3.32]
  Serotype 23F: number analyzed (Participants) | 175 | 81
  Serotype 23F | 2.05 [1.79 to 2.34] | 1.61 [1.38 to 1.88]

8. Secondary Outcome: Percentage of Participants With Anti-pneumococcal Antibody Concentrations (>=0.35 mcg/mL and >=1.0 mcg/mL) After Prevnar 13® Vaccine Administered Alone or Along With MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2 (up to the Infant Age of 6 Months)
Description: Percentage of participants with anti-pneumococcal antibody concentrations >=0.35 micrograms per milliliter (mcg/mL) and >=1.0 mcg/mL for Prevnar 13 serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F was reported in this outcome measure. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: as for outcome 7
Population: Analysis was performed on PPAS1. Here, 'Number analyzed'=participants with available data for specified categories. Data for this outcome measure was not planned to be collected and analyzed for Groups 3 and 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 2: Menveo® Vaccine (Mexico): Participants aged 2 months (at the time of enrollment) received Menveo® vaccine at the age of Months 2, 4, 6, and 12 along with Prevnar 13®, Hexacima®, vaccines at the age of Months 2, 4, 6 and 12; RotaTeq® vaccine at the age of Months 2, 4 and 6 and MMR®II vaccine at the age of Month 12.
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 176 | 81
percentage of participants
  Serotype 1: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 1: >=0.35 mcg/mL | 100 [97.9 to 100] | 100 [95.5 to 100]
  Serotype 3: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 3: >=0.35 mcg/mL | 81.7 [75.2 to 87.1] | 74.1 [63.1 to 83.2]
  Serotype 4: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 4: >=0.35 mcg/mL | 99.4 [96.9 to 100] | 98.8 [93.3 to 100]
  Serotype 5: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 5: >=0.35 mcg/mL | 99.4 [96.9 to 100] | 100 [95.5 to 100]
  Serotype 6A: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 6A: >=0.35 mcg/mL | 100 [97.9 to 100] | 100 [95.5 to 100]
  Serotype 6B: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 6B: >=0.35 mcg/mL | 97.7 [94.3 to 99.4] | 98.8 [93.3 to 100]
  Serotype 7F: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 7F: >=0.35 mcg/mL | 100 [97.9 to 100] | 100 [95.5 to 100]
  Serotype 9V: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 9V: >=0.35 mcg/mL | 100 [97.9 to 100] | 100 [95.5 to 100]
  Serotype 14: >=0.35 mcg/mL: number analyzed (Participants) | 174 | 81
  Serotype 14: >=0.35 mcg/mL | 100 [97.9 to 100] | 100 [95.5 to 100]
  Serotype 18C: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 18C: >=0.35 mcg/mL | 100 [97.9 to 100] | 97.5 [91.4 to 99.7]
  Serotype 19A: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 19A: >=0.35 mcg/mL | 99.4 [96.9 to 100] | 100 [95.5 to 100]
  Serotype 19F: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 19F: >=0.35 mcg/mL | 99.4 [96.9 to 100] | 98.8 [93.3 to 100]
  Serotype 23F: >=0.35 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 23F: >=0.35 mcg/mL | 96.0 [91.9 to 98.4] | 96.3 [89.6 to 99.2]
  Serotype 1: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 1: >=1.0 mcg/mL | 95.4 [91.2 to 98.0] | 95.1 [87.8 to 98.6]
  Serotype 3: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 3: >=1.0 mcg/mL | 20.0 [14.3 to 26.7] | 14.8 [7.9 to 24.4]
  Serotype 4: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 4: >=1.0 mcg/mL | 84.0 [77.7 to 89.1] | 79.0 [68.5 to 87.3]
  Serotype 5: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 5: >=1.0 mcg/mL | 88.6 [82.9 to 92.9] | 81.5 [71.3 to 89.2]
  Serotype 6A: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 6A: >=1.0 mcg/mL | 96.6 [92.7 to 98.7] | 96.3 [89.6 to 99.2]
  Serotype 6B: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 6B: >=1.0 mcg/mL | 88.6 [82.9 to 92.9] | 81.5 [71.3 to 89.2]
  Serotype 7F: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 7F: >=1.0 mcg/mL | 99.4 [96.9 to 100] | 100 [95.5 to 100]
  Serotype 9V: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 9V: >=1.0 mcg/mL | 86.9 [80.9 to 91.5] | 85.2 [75.6 to 92.1]
  Serotype 14: >=1.0 mcg/mL: number analyzed (Participants) | 174 | 81
  Serotype 14: >=1.0 mcg/mL | 98.9 [95.9 to 99.9] | 100 [95.5 to 100]
  Serotype 18C: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 18C: >=1.0 mcg/mL | 90.9 [85.6 to 94.7] | 81.5 [71.3 to 89.2]
  Serotype 19A: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 19A: >=1.0 mcg/mL | 86.9 [80.9 to 91.5] | 84.0 [74.1 to 91.2]
  Serotype 19F: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 19F: >=1.0 mcg/mL | 97.7 [94.3 to 99.4] | 98.8 [93.3 to 100]
  Serotype 23F: >=1.0 mcg/mL: number analyzed (Participants) | 175 | 81
  Serotype 23F: >=1.0 mcg/mL | 81.1 [74.5 to 86.6] | 79.0 [68.5 to 87.3]

9. Secondary Outcome: Percentage of Participants With >=3-fold and >=4-fold Rise in Anti-rotavirus Serum IgA Antibody Concentrations After RotaTeq® Vaccine Administered Alone or Along With MenACYW Conjugate or Menveo® Vaccine: Groups 1 & 2 (up to the Infant Age of 6 Months)
Description: Anti-rotavirus IgA antibodies in human serum was measured by ELISA. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days after 6-months vaccination) to pre-dose titer at age of 2 months (i.e., Day 0). Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: From Day 0 (before the first vaccination with RotaTeq® vaccine at the age of 2 months), 30 days after the vaccination with RotaTeq® vaccine at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 176 | 81
percentage of participants
  >=3-fold rise | 93.8 [89.1 to 96.8] | 91.4 [83.0 to 96.5]
  >=4-fold rise | 93.8 [89.1 to 96.8] | 88.9 [80.0 to 94.8]

10. Secondary Outcome: Geometric Mean Titers (GMTs) of MMR Antibodies Following Vaccination With M-M-R®II Vaccine Administered Alone or Along With the MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2
Description: GMTs against anti-measles and anti-rubella antibodies were measured by Bulk Measles immunoglobulin G (IgG) Enzyme Immunoassay (EIA) and anti-mumps antibodies were assessed by ELISA. Titers were expressed in terms of 1/dilution.
Time Frame: 30 days after the vaccination with M-M-R®II vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure and 'Number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 125 | 60
titers
  Anti-Measles | 5256 [4718 to 5855] | 5679 [5120 to 6299]
  Anti-Mumps: number analyzed (Participants) | 125 | 59
  Anti-Mumps | 130 [114 to 149] | 109 [83.7 to 142]
  Anti-Rubella | 117 [104 to 132] | 117 [100 to 136]

11. Secondary Outcome: Geometric Mean Concentration of Anti-pneumococcal Antibodies Following Vaccination With Prevnar 13® Vaccine Administered Alone or Along With the MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2
Description: GMCs against Streptococcus pneumoniae polysaccharide (PS) serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F were measured by ECL assay. Concentration was expressed in terms of titers (1/dilution).
Time Frame: 30 days after the vaccination with Prevnar13® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Groups 3 and 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 125 | 60
titers
  Serotype 1 | 2.96 [2.49 to 3.52] | 2.74 [2.10 to 3.57]
  Serotype 3 | 0.504 [0.431 to 0.590] | 0.518 [0.398 to 0.674]
  Serotype 4 | 1.59 [1.32 to 1.93] | 1.36 [1.04 to 1.79]
  Serotype 5 | 2.48 [2.09 to 2.95] | 2.18 [1.73 to 2.74]
  Serotype 6A | 7.22 [5.92 to 8.80] | 5.85 [4.33 to 7.91]
  Serotype 6B | 4.89 [3.96 to 6.03] | 4.06 [3.03 to 5.46]
  Serotype 7F | 3.79 [3.21 to 4.48] | 3.91 [3.12 to 4.91]
  Serotype 9V | 2.59 [2.14 to 3.14] | 2.31 [1.76 to 3.03]
  Serotype 14 | 7.55 [6.18 to 9.22] | 7.47 [5.72 to 9.74]
  Serotype 18C | 2.35 [1.97 to 2.82] | 1.79 [1.35 to 2.39]
  Serotype 19A | 4.13 [3.35 to 5.09] | 4.18 [3.16 to 5.53]
  Serotype 19F | 4.15 [3.41 to 5.05] | 3.84 [2.80 to 5.25]
  Serotype 23F | 3.13 [2.52 to 3.90] | 2.53 [1.80 to 3.56]

12. Secondary Outcome: Percentage of Participants With Anti-pneumococcal Antibody Concentrations (>=0.35 mcg/mL and >=1.0 mcg/mL) Following Vaccination With Prevnar13® Vaccine Administered Alone or Along With the MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2
Description: Percentage of participants with anti-pneumococcal antibody concentrations >=0.35 mcg/mL and >=1.0 mcg/mL for Prevnar 13 serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F was reported in this outcome measure.
Time Frame: 30 days after the vaccination with Prevnar 13® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Here, "overall number of participants analyzed" = participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Groups 3 and 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 125 | 60
percentage of participants
  Serotype 1: >=0.35 mcg/mL | 97.6 [93.1 to 99.5] | 98.3 [91.1 to 100]
  Serotype 3: >=0.35 mcg/mL | 68.8 [59.9 to 76.8] | 66.7 [53.3 to 78.3]
  Serotype 4: >=0.35 mcg/mL | 90.4 [83.8 to 94.9] | 86.7 [75.4 to 94.1]
  Serotype 5: >=0.35 mcg/mL | 95.2 [89.8 to 98.2] | 96.7 [88.5 to 99.6]
  Serotype 6A: >=0.35 mcg/mL | 98.4 [94.3 to 99.8] | 100 [94.0 to 100]
  Serotype 6B: >=0.35 mcg/mL | 95.2 [89.8 to 98.2] | 93.3 [83.8 to 98.2]
  Serotype 7F: >=0.35 mcg/mL | 99.2 [95.6 to 100] | 100 [94.0 to 100]
  Serotype 9V: >=0.35 mcg/mL | 93.6 [87.8 to 97.2] | 90.0 [79.5 to 96.2]
  Serotype 14: >=0.35 mcg/mL | 99.2 [95.6 to 100] | 98.3 [91.1 to 100]
  Serotype 18C: >=0.35 mcg/mL | 93.6 [87.8 to 97.2] | 85.0 [73.4 to 92.9]
  Serotype 19A: >=0.35 mcg/mL | 96.0 [90.9 to 98.7] | 100 [94.0 to 100]
  Serotype 19F: >=0.35 mcg/mL | 97.6 [93.1 to 99.5] | 91.7 [81.6 to 97.2]
  Serotype 23F: >=0.35 mcg/mL | 93.6 [87.8 to 97.2] | 90.0 [79.5 to 96.2]
  Serotype 1: >=1.0 mcg/mL | 84.0 [76.4 to 89.9] | 80.0 [67.7 to 89.2]
  Serotype 3: >=1.0 mcg/mL | 20.0 [13.4 to 28.1] | 25.0 [14.7 to 37.9]
  Serotype 4: >=1.0 mcg/mL | 72.0 [63.3 to 79.7] | 65.0 [51.6 to 76.9]
  Serotype 5: >=1.0 mcg/mL | 84.8 [77.3 to 90.6] | 81.7 [69.6 to 90.5]
  Serotype 6A: >=1.0 mcg/mL | 90.4 [83.8 to 94.9] | 86.7 [75.4 to 94.1]
  Serotype 6B: >=1.0 mcg/mL | 88.8 [81.9 to 93.7] | 86.7 [75.4 to 94.1]
  Serotype 7F: >=1.0 mcg/mL | 90.4 [83.8 to 94.9] | 90.0 [79.5 to 96.2]
  Serotype 9V: >=1.0 mcg/mL | 80.8 [72.8 to 87.3] | 80.0 [67.7 to 89.2]
  Serotype 14: >=1.0 mcg/mL | 94.4 [88.8 to 97.7] | 96.7 [88.5 to 99.6]
  Serotype 18C: >=1.0 mcg/mL | 82.4 [74.6 to 88.6] | 78.3 [65.8 to 87.9]
  Serotype 19A: >=1.0 mcg/mL | 84.0 [76.4 to 89.9] | 85.0 [73.4 to 92.9]
  Serotype 19F: >=1.0 mcg/mL | 84.8 [77.3 to 90.6] | 83.3 [71.5 to 91.7]
  Serotype 23F: >=1.0 mcg/mL | 82.4 [74.6 to 88.6] | 80.0 [67.7 to 89.2]

13. Secondary Outcome: Percentage of Participants With Anti-MMR Antibodies (Ab) Concentrations Following Vaccination With MMR Vaccine Administered Alone or Along With the MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2
Description: Percentage of participants with anti-measles Ab concentrations >=255 milli-international unit per milliliter (mIU/mL), anti-mumps Ab concentrations: >=10 Ab units/mL, and anti-rubella Ab concentrations >=10 international unit per milliliter (IU/mL) was reported in this outcome measure.
Time Frame: 30 days after the vaccination with M-M-R®II vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Here, "overall number of participants analyzed" = participants with available data for this outcome measure and 'Number analyzed'=participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 125 | 60
percentage of participants
  Anti-Measles | 99.2 [95.6 to 100] | 100 [94.0 to 100]
  Anti-Mumps: number analyzed (Participants) | 125 | 59
  Anti-Mumps | 100 [97.1 to 100] | 96.6 [88.3 to 99.6]
  Anti-Rubella | 100 [97.1 to 100] | 100 [94.0 to 100]

14. Secondary Outcome: Percentage of Participants With Antibodies Concentrations Following Vaccination With Hexacima® (DTaP-IPV-HB-Hib) Vaccine Administered Alone or Along With the MenACYW Conjugate Vaccine: Groups 1 and 2
Description: Percentage of participants with anti-diphtheria Ab concentrations: >= 0.1 and 1 IU/mL, and anti-tetanus Ab concentrations: >= 0.1 and 1 IU/mL, anti-poliovirus types 1, 2, and 3 Ab titers >= 8 (1/dilution), anti-hepatitis B surface (HBs) antigen Ab concentrations: >= 10 and >= 100 mIU/mL and anti-polyribosyl-ribitol phosphate (anti-PRP) Ab concentrations: >= 0.15 and 1.0 microgram per milliliter (mcg/mL) was reported in this outcome measure.
Time Frame: 30 days after the vaccination with Hexacima® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Groups 3 and 4. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 125 | 60
percentage of participants
  Anti-Diphtheria: >=0.1 | 100 [97.1 to 100] | 100 [94.0 to 100]
  Anti-Diphtheria: >=1 | 98.4 [94.3 to 99.8] | 93.3 [83.8 to 98.2]
  Anti-Tetanus: >=0.1 | 100 [97.1 to 100] | 100 [94.0 to 100]
  Anti-Tetanus: >=1 | 100 [97.1 to 100] | 98.3 [91.1 to 100]
  Anti-Polio 1: >=8 | 100 [97.1 to 100] | 100 [94.0 to 100]
  Anti-Polio 2: >=8 | 100 [97.1 to 100] | 100 [94.0 to 100]
  Anti-Polio 3: >=8 | 100 [97.1 to 100] | 100 [94.0 to 100]
  Anti-Hepatitis B: >=10 | 100 [97.1 to 100] | 100 [94.0 to 100]
  Anti-Hepatitis B: >=100 | 100 [97.1 to 100] | 100 [94.0 to 100]
  Anti-PRP: >=0.15 | 100 [97.1 to 100] | 98.3 [91.1 to 100]
  Anti-PRP: >=1.0 | 100 [97.1 to 100] | 98.3 [91.1 to 100]

15. Secondary Outcome: Percentage of Participants With Vaccine Response for Pertussis (PT) and FHA Antibodies Following Vaccination With Hexacima® (DTaP-IPV-HB-Hib) Vaccine Administered Alone or Along With the MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2
Description: Pertussis and FHA vaccine response was defined as: if the pre-vaccination concentration was >=4*lower limit of quantification (LLOQ), then the post-vaccination concentration was >=pre-vaccination concentration and if the pre-vaccination concentration was <4*LLOQ, then the post-booster vaccination concentration was >= 4*LLOQ. The LLOQ was equal to 2.00 Endotoxin units per milliliter (EU/mL).
Time Frame: 30 days after the vaccination with Hexacima® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Here, "overall number of participants analyzed" = participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 125 | 60
percentage of participants
  PT | 92.8 [86.8 to 96.7] | 95.0 [86.1 to 99.0]
  FHA | 91.2 [84.8 to 95.5] | 83.3 [71.5 to 91.7]

16. Secondary Outcome: Geometric Mean Concentration of PT and FHA Antibodies Before Vaccination With Pentaxim® (DTaP-Hib-IPV) Vaccine Administered Alone or Along With the MenACYW Conjugate Vaccine: Groups 3 and 4 (up to the Infant Age of 6 Months)
Description: GMCs for PT and FHA were measured by ECL assay. Concentration was expressed in terms of titers (1/dilution). Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: Day 0 (before first vaccination with Pentaxim® vaccine) of the infant series (i.e., at the age of 2 months)
Population: Analysis was performed on PPAS1. Here, "overall number of participants analyzed" = participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Groups 1 and 2.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 96 | 53
titers
  PT | 2.03 [1.64 to 2.51] | 1.75 [1.35 to 2.25]
  FHA | 6.99 [5.53 to 8.84] | 6.23 [4.36 to 8.88]

17. Secondary Outcome: Percentage of Participants With Antibodies Concentrations Following Vaccination With Pentaxim® (DTaP-Hib-IPV) Vaccine Administered Alone or Along With the MenACYW Conjugate Vaccine: Groups 3 and 4 (up to the Infant Age of 6 Months)
Description: Percentage of participants with anti-diphtheria Ab concentrations: >= 0.1 and 1 IU/mL, anti-tetanus Ab concentrations: >= 0.1 and 1 IU/mL, anti-poliovirus types 1, 2, and 3 Ab titers >= 8 (1/dilution), and anti-PRP Ab concentrations: >= 0.15 and 1.0 mcg/mL were reported in this outcome measure. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the vaccination with Pentaxim® vaccine at the age of 6 months of the infant series (i.e., at the age of Month 7)
Population: Analysis was performed on PPAS1. Here, 'Number analyzed'=participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Groups 1 and 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 97 | 53
percentage of participants
  Anti-Diphtheria: >=0.1: number analyzed (Participants) | 95 | 53
  Anti-Diphtheria: >=0.1 | 98.9 [94.3 to 100] | 92.5 [81.8 to 97.9]
  Anti-Diphtheria: >=1: number analyzed (Participants) | 95 | 53
  Anti-Diphtheria: >=1 | 80.0 [70.5 to 87.5] | 71.7 [57.7 to 83.2]
  Anti-Tetanus: >=0.1: number analyzed (Participants) | 95 | 53
  Anti-Tetanus: >=0.1 | 100 [96.2 to 100] | 98.1 [89.9 to 100]
  Anti-Tetanus: >=1: number analyzed (Participants) | 95 | 53
  Anti-Tetanus: >=1 | 74.7 [64.8 to 83.1] | 54.7 [40.4 to 68.4]
  Anti-Polio 1: >=8: number analyzed (Participants) | 89 | 47
  Anti-Polio 1: >=8 | 100 [95.9 to 100] | 100 [92.5 to 100]
  Anti-Polio 2: >=8: number analyzed (Participants) | 89 | 47
  Anti-Polio 2: >=8 | 100 [95.9 to 100] | 100 [92.5 to 100]
  Anti-Polio 3: >=8: number analyzed (Participants) | 89 | 47
  Anti-Polio 3: >=8 | 100 [95.9 to 100] | 100 [92.5 to 100]
  Anti-PRP: >=0.15: number analyzed (Participants) | 90 | 52
  Anti-PRP: >=0.15 | 94.4 [87.5 to 98.2] | 90.4 [79.0 to 96.8]
  Anti-PRP: >=1.0: number analyzed (Participants) | 90 | 52
  Anti-PRP: >=1.0 | 72.2 [61.8 to 81.1] | 57.7 [43.2 to 71.3]

18. Secondary Outcome: Percentage of Participants With Vaccine Response for PT and FHA Antibodies Following Vaccination With Pentaxim® (DTaP-Hib-IPV) Vaccine Administered Alone or Along With the MenACYW Conjugate Vaccine: Groups 3 and 4 (up to the Infant Age of 6 Months)
Description: Pertussis and FHA vaccine response was defined as: if the pre-vaccination concentration was >=4*LLOQ, then the post-vaccination concentration was >= pre-vaccination concentration and if the pre-vaccination concentration was <4*LLOQ, then the post-booster vaccination concentration was >= 4*LLOQ. The LLOQ was equal to 2.00 EU/mL. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the vaccination with Pentaxim® vaccine at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Here, "overall number of participants analyzed" = participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 94 | 53
percentage of participants
  PT | 97.9 [92.5 to 99.7] | 90.6 [79.3 to 96.9]
  FHA | 97.9 [92.5 to 99.7] | 94.3 [84.3 to 98.8]

19. Secondary Outcome: Percentage of Participants With Anti-Hepatitis (HBs) Concentrations Following Vaccination With ENGERIX-B® (Hepatitis B) Vaccine Administered Alone or Along With the MenACYW Conjugate Vaccine: Groups 3 and 4 (up to the Infant Age of 6 Months)
Description: Percentage of participants with anti-hepatitis B surface (HBs) antigen Ab concentrations: >=10 and >=100 mIU/mL was presented in this outcome measure. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the vaccination with ENGERIX-B® vaccine at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 87 | 50
percentage of participants
  Anti-HBs: >=10 | 97.7 [91.9 to 99.7] | 98.0 [89.4 to 99.9]
  Anti-HBs: >=100 | 93.1 [85.6 to 97.4] | 80.0 [66.3 to 90.0]

20. Secondary Outcome: Geometric Mean Concentrations of MMR Antibodies Following Vaccination With MMR Vaccine Administered Alone or Along With the MenACYW Conjugate Vaccine: Groups 3 and 4
Description: GMCs against anti-measles and anti-rubella antibodies were measured by Bulk Measles IgG EIA, and anti-mumps antibodies were assessed by ELISA. Concentrations were expressed in terms of titers (1/dilution).
Time Frame: 30 days after the vaccination with MMR vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 96 | 50
titers
  Anti-Measles | 1461 [1128 to 1893] | 1233 [800 to 1901]
  Anti-Mumps | 50.5 [40.4 to 63.1] | 53.5 [40.8 to 70.2]
  Anti-Rubella | 47.6 [39.5 to 57.2] | 55.2 [42.3 to 72.1]

21. Secondary Outcome: Percentage of Participants With Anti-MMR Concentrations Following Vaccination With MMR Vaccine Administered Alone or Along With the MenACYW Vaccine or Routine Pediatric Vaccines: Groups 3 and 4
Description: Percentage of participants with anti-measles Ab concentrations >=255 mIU/mL, anti-mumps Ab concentrations: >=10 Ab units/mL, and anti-rubella Ab concentrations >=10 IU/mL was reported in this outcome measure.
Time Frame: 30 days after the vaccination with MMR vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 96 | 50
percentage of participants
  Anti-Measles | 93.8 [86.9 to 97.7] | 88.0 [75.7 to 95.5]
  Anti-Mumps | 89.6 [81.7 to 94.9] | 90.0 [78.2 to 96.7]
  Anti-Rubella | 95.8 [89.7 to 98.9] | 94.0 [83.5 to 98.7]

22. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA Before Vaccination With MenACYW Conjugate or Menveo® Vaccine: Groups 1, 2 and 3 (up to the Infant Age of 6 Months)
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: Day 0 (before the first vaccination with MenACYW Conjugate or Menveo® Vaccine) of the infant series (i.e., at the age of 2 months)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 176 | 81 | 97
titers
  Serogroup A | 2.65 [2.39 to 2.93] | 2.24 [2.10 to 2.38] | 2.88 [2.64 to 3.14]
  Serogroup C | 2.16 [2.08 to 2.23] | 2.29 [2.13 to 2.47] | 2.16 [2.04 to 2.30]
  Serogroup Y | 2.62 [2.45 to 2.81] | 2.89 [2.51 to 3.33] | 2.37 [2.07 to 2.72]
  Serogroup W | 3.57 [3.21 to 3.97] | 3.15 [2.79 to 3.55] | 2.18 [2.04 to 2.32]

23. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA Following MenACYW Conjugate Vaccine: Groups 1 and 3 (up to the Infant Age of 6 Months)
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution. Group 2 data were presented separately. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the vaccination with MenACYW Conjugate vaccine at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 176 | 97
titers
  Serogroup A | 71.7 [56.8 to 90.7] | 31.5 [22.2 to 44.9]
  Serogroup C | 626 [549 to 714] | 267 [196 to 365]
  Serogroup Y | 246 [216 to 281] | 78.2 [60.3 to 101]
  Serogroup W | 340 [294 to 393] | 78.7 [61.9 to 100]

24. Secondary Outcome: Percentage of Participants With Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccines: Groups 1 and 3 (up to the Infant Age of 6 Months)
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Group 2 data were presented separately. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the vaccination with MenACYW Conjugate vaccine at the age of 6 months of the infant series (i.e., at the age of Month 7)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 176 | 97
percentage of participants
  Serogroup A: >=1:4 | 96.0 [92.0 to 98.4] | 93.8 [87.0 to 97.7]
  Serogroup A: >=1:8 | 90.9 [85.7 to 94.7] | 78.4 [68.8 to 86.1]
  Serogroup C: >=1:4 | 100 [97.9 to 100] | 94.8 [88.4 to 98.3]
  Serogroup C: >=1:8 | 100 [97.9 to 100] | 94.8 [88.4 to 98.3]
  Serogroup Y: >=1:4 | 99.4 [96.9 to 100] | 94.8 [88.4 to 98.3]
  Serogroup Y: >=1:8 | 99.4 [96.9 to 100] | 92.8 [85.7 to 97.0]
  Serogroup W: >=1:4 | 99.4 [96.9 to 100] | 94.8 [88.4 to 98.3]
  Serogroup W: >=1:8 | 99.4 [96.9 to 100] | 94.8 [88.4 to 98.3]

25. Secondary Outcome: Percentage of Participants With >=4-Fold Rise in Antibody Titers Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine: Groups 1 and 3 (up to the Infant Age of 6 Months)
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days after the 6-months vaccination) to pre-dose titer at 2 months of age (i.e., Day 0). Group 2 data were presented separately. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: From Day 0 (before the first vaccination, at the age of 2 months), 30 days after vaccination with MenACYW Conjugate vaccine at the age of 6 months of infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 176 | 97
percentage of participants
  Serogroup A | 84.7 [78.5 to 89.6] | 70.1 [60.0 to 79.0]
  Serogroup C | 100 [97.9 to 100] | 94.8 [88.4 to 98.3]
  Serogroup Y | 99.4 [96.9 to 100] | 87.6 [79.4 to 93.4]
  Serogroup W | 98.3 [95.1 to 99.6] | 93.8 [87.0 to 97.7]

26. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA Following Vaccination With Menveo® Vaccine: Group 2 (up to the Infant Age of 6 Months)
Description: as for outcome 22
Time Frame: 30 days after the vaccination with Menveo® vaccine at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 81
titers
  Serogroup A | 16.7 [12.0 to 23.3]
  Serogroup C | 62.4 [47.2 to 82.4]
  Serogroup Y | 59.8 [46.9 to 76.1]
  Serogroup W | 95.7 [78.4 to 117]

27. Secondary Outcome: Percentage of Participants With Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With Menveo® Vaccine: Group 2 (up to the Infant Age of 6 Months)
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: as for outcome 26
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 81
percentage of participants
  Serogroup A: >=1:4 | 85.2 [75.6 to 92.1]
  Serogroup A: >=1:8 | 69.1 [57.9 to 78.9]
  Serogroup C: >=1:4 | 98.8 [93.3 to 100]
  Serogroup C: >=1:8 | 97.5 [91.4 to 99.7]
  Serogroup Y: >=1:4 | 98.8 [93.3 to 100]
  Serogroup Y: >=1:8 | 97.5 [91.4 to 99.7]
  Serogroup W: >=1:4 | 100 [95.5 to 100]
  Serogroup W: >=1:8 | 100 [95.5 to 100]

28. Secondary Outcome: Percentage of Participants With >=4-Fold Rise in Antibody Titers Against Meningococcal Serogroups A, C, Y, and W Following Vaccinations With Menveo® Vaccine: Group 2 (up to the Infant Age of 6 Months)
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days after the vaccination at the age of 6 months) to pre-dose titer at Day 0 (i.e., before the first vaccination, at 2 months of age). Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: Day 0 (before the first vaccination, at the age of 2 months), 30 days after vaccination with Menveo® vaccines at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 81
percentage of participants
  Serogroup A | 58.0 [46.5 to 68.9]
  Serogroup C | 86.4 [77.0 to 93.0]
  Serogroup Y | 92.6 [84.6 to 97.2]
  Serogroup W | 97.5 [91.4 to 99.7]

29. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA Antibodies Following Last Vaccination With MenACYW Conjugate Vaccine: Groups 1 and 3
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution. Group 2 data were presented separately.
Time Frame: 30 days after the vaccination with MenACYW Conjugate vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Group 4. Here, 'Number analyzed'=participants with available data for the specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Group 1: MenACYW Conjugate Vaccine (Mexico): Participants aged 2 months (at the time of enrollment) received MenACYW Conjugate vaccine at the age of Months 2, 6, and 12 along with Prevnar 13®, Hexacima® vaccines at the age of Months 2, 4, 6 and 12; RotaTeq® vaccine at the age of Months 2, 4 and 6, and MMR®II vaccine at the age of Month 12.
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 126 | 96
titers
  Serogroup A | 145 [114 to 185] | 85.4 [54.0 to 135]
  Serogroup C | 897 [742 to 1086] | 214 [130 to 353]
  Serogroup Y: number analyzed (Participants) | 125 | 96
  Serogroup Y | 401 [343 to 469] | 97.3 [63.4 to 149]
  Serogroup W: number analyzed (Participants) | 125 | 96
  Serogroup W | 639 [542 to 754] | 123 [77.1 to 195]

30. Secondary Outcome: Percentage of Participants With Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine: Groups 1 and 3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Group 2 data were presented separately.
Time Frame: 30 days after the vaccination with MenACYW Conjugate vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Group 4. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 126 | 96
percentage of participants
  Serogroup A: >=1:4 | 98.4 [94.4 to 99.8] | 97.9 [92.7 to 99.7]
  Serogroup A: >=1:8 | 97.6 [93.2 to 99.5] | 89.6 [81.7 to 94.9]
  Serogroup C: >=1:4 | 100 [97.1 to 100] | 91.7 [84.2 to 96.3]
  Serogroup C: >=1:8 | 99.2 [95.7 to 100] | 82.3 [73.2 to 89.3]
  Serogroup Y: >=1:4: number analyzed (Participants) | 125 | 96
  Serogroup Y: >=1:4 | 100 [97.1 to 100] | 83.3 [74.4 to 90.2]
  Serogroup Y: >=1:8: number analyzed (Participants) | 125 | 96
  Serogroup Y: >=1:8 | 100 [97.1 to 100] | 80.2 [70.8 to 87.6]
  Serogroup W: >=1:4: number analyzed (Participants) | 125 | 96
  Serogroup W: >=1:4 | 100 [97.1 to 100] | 85.4 [76.7 to 91.8]
  Serogroup W: >=1:8: number analyzed (Participants) | 125 | 96
  Serogroup W: >=1:8 | 100 [97.1 to 100] | 80.2 [70.8 to 87.6]

31. Secondary Outcome: Percentage of Participants With >=4-Fold Rise in Antibody Titers Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine: Groups 1 and 3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days after the vaccination at the age of 6 months) to pre-dose titer at Day 0 (i.e., before the first vaccination, at the age of 2 months). Group 2 data were presented separately.
Time Frame: Day 0 (before the first vaccination, at the age of 2 months), 30 days after the vaccination with MenACYW Conjugate vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Here, 'Number analyzed'=participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 126 | 96
percentage of participants
  Serogroup A | 96.8 [92.1 to 99.1] | 74.0 [64.0 to 82.4]
  Serogroup C | 99.2 [95.7 to 100] | 81.3 [72.0 to 88.5]
  Serogroup Y: number analyzed (Participants) | 125 | 96
  Serogroup Y | 100 [97.1 to 100] | 80.2 [70.8 to 87.6]
  Serogroup W: number analyzed (Participants) | 125 | 96
  Serogroup W | 99.2 [95.6 to 100] | 79.2 [69.7 to 86.8]

32. Secondary Outcome: Percentage of Participants Achieving Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W Following Last Vaccination With MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 3
Description: The hSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination hSBA titer >=1:16 for participants with pre-vaccination hSBA titer <1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >=1:8. Group 2 data were presented separately.
Time Frame: 30 days after the vaccination with MenACYW Conjugate vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Here, 'Number analyzed'=participants with available data for specified categories. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 126 | 96
percentage of participants
  Serogroup A | 96.8 [92.1 to 99.1] | 74.0 [64.0 to 82.4]
  Serogroup C | 99.2 [95.7 to 100] | 81.3 [72.0 to 88.5]
  Serogroup Y: number analyzed (Participants) | 125 | 96
  Serogroup Y | 100 [97.1 to 100] | 80.2 [70.8 to 87.6]
  Serogroup W: number analyzed (Participants) | 125 | 96
  Serogroup W | 99.2 [95.6 to 100] | 79.2 [69.7 to 86.8]

33. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA Antibodies Following Last Vaccination With Menveo® Vaccine: Group 2
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: 30 days after the vaccination with Menveo® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 60
titers
  Serogroup A | 65.5 [44.5 to 96.3]
  Serogroup C | 77.0 [52.5 to 113]
  Serogroup Y | 228 [173 to 301]
  Serogroup W | 242 [184 to 318]

34. Secondary Outcome: Percentage of Participants With Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With Menveo® Vaccine: Group 2
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay.
Time Frame: 30 days after the vaccination with Menveo® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 60
percentage of participants
  Serogroup A: >=1:4 | 96.7 [88.5 to 99.6]
  Serogroup A: >=1:8 | 95.0 [86.1 to 99.0]
  Serogroup C: >=1:4 | 96.7 [88.5 to 99.6]
  Serogroup C: >=1:8 | 93.3 [83.8 to 98.2]
  Serogroup Y: >=1:4 | 100 [94.0 to 100]
  Serogroup Y: >=1:8 | 100 [94.0 to 100]
  Serogroup W: >=1:4 | 100 [94.0 to 100]
  Serogroup W: >=1:8 | 100 [94.0 to 100]

35. Secondary Outcome: Percentage of Participants With >=4-Fold Rise in Antibody Titers Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With Menveo® Vaccine: Group 2
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Fold-rise was calculated as ratio of post-vaccination titer (i.e., 30 days after the vaccination at the age of 12 months) to pre-dose titer at Day 0 (i.e., before first vaccination, at the age of 2 months).
Time Frame: Day 0 (before the first vaccination, at the age of Month 2), 30 days after the vaccination with Menveo® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 60
percentage of participants
  Serogroup A | 85.0 [73.4 to 92.9]
  Serogroup C | 88.3 [77.4 to 95.2]
  Serogroup Y | 96.7 [88.5 to 99.6]
  Serogroup W | 100 [94.0 to 100]

36. Secondary Outcome: Percentage of Participants Achieving Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W Following Last Vaccination With Menveo® Vaccine: Group 2
Description: The hSBA vaccine seroresponse against serogroups A, C, Y, and W was defined as post-vaccination hSBA titer >=1:16 for participants with pre-vaccination hSBA titer <1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >=1:8.
Time Frame: 30 days after the vaccination with Menveo® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 60
percentage of participants
  Serogroup A | 85.0 [73.4 to 92.9]
  Serogroup C | 88.3 [77.4 to 95.2]
  Serogroup Y | 96.7 [88.5 to 99.6]
  Serogroup W | 100 [94.0 to 100]

37. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by Serum Bactericidal Assay Using Baby Rabbit Complement Following MenACYW Conjugate or Menveo® Vaccine: Groups 1 and 2 (up to the Infant Age of 6 Months)
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by serum bactericidal assay using rabbit complement (rSBA). Titers were expressed in terms of 1/dilution. Group 3 data were presented separately. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: Day 0 (before the first vaccination, at the age of 2 months), 30 days after the vaccination with MenACYW Conjugate vaccine at the age of 6 months (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Here, "overall number of participants analyzed" = participants with available data for this outcome measure and 'Number analyzed'=participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 90 | 40
titers
  Serogroup A: Day 0 | 2.09 [1.96 to 2.23] | 2.03 [1.96 to 2.11]
  Serogroup A: 30 days post-vaccination: number analyzed (Participants) | 89 | 40
  Serogroup A: 30 days post-vaccination | 387 [293 to 510] | 1328 [708 to 2489]
  Serogroup C: Day 0 | 2.05 [1.95 to 2.14] | 2.38 [1.85 to 3.05]
  Serogroup C: 30 days post-vaccination: number analyzed (Participants) | 89 | 40
  Serogroup C: 30 days post-vaccination | 1366 [1138 to 1640] | 235 [173 to 319]
  Serogroup Y: Day 0 | 2.28 [1.93 to 2.69] | 2.93 [1.89 to 4.54]
  Serogroup Y: 30 days post-vaccination: number analyzed (Participants) | 89 | 40
  Serogroup Y: 30 days post-vaccination | 1056 [872 to 1280] | 549 [336 to 897]
  Serogroup W: Day 0 | 2.00 [NA to NA] — The 95% confidence interval was not computed as the standard deviation of the sample was 0, since all participants had the same value. | 2.00 [NA to NA] — The 95% confidence interval was not computed as the standard deviation of the sample was 0, since all participants had the same value.
  Serogroup W: 30 days post-vaccination: number analyzed (Participants) | 89 | 40
  Serogroup W: 30 days post-vaccination | 2587 [2071 to 3231] | 763 [509 to 1143]

38. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by rSBA Following MenACYW Conjugate Vaccine: Group 3 (up to the Infant Age of 6 Months)
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by serum bactericidal assay using rabbit complement (rSBA). Titers were expressed in terms of 1/dilution. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: Day 0 (before the first vaccination, at the age of Month 2), 30 days after the vaccination of MenACYW Conjugate vaccine at the age of 6 months (i.e., at the age of 7 months)
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 56
titers
  Serogroup A: Day 0: number analyzed (Participants) | 55
  Serogroup A: Day 0 | 2.18 [1.83 to 2.61]
  Serogroup A: 30 days post-vaccination: number analyzed (Participants) | 41
  Serogroup A: 30 days post-vaccination | 213 [126 to 358]
  Serogroup C: Day 0 | 2.02 [1.98 to 2.08]
  Serogroup C: 30 days post-vaccination: number analyzed (Participants) | 45
  Serogroup C: 30 days post-vaccination | 460 [286 to 738]
  Serogroup Y: Day 0 | 2.15 [1.86 to 2.50]
  Serogroup Y: 30 days post-vaccination: number analyzed (Participants) | 43
  Serogroup Y: 30 days post-vaccination | 817 [587 to 1138]
  Serogroup W: Day 0 | 2.15 [1.93 to 2.40]
  Serogroup W: 30 days post-vaccination: number analyzed (Participants) | 44
  Serogroup W: 30 days post-vaccination | 961 [593 to 1558]

39. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by rSBA Following Last Vaccination With MenACYW Conjugate Vaccine or Menveo® Vaccine: Groups 1 and 2
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by rSBA. Titers were expressed in terms of 1/dilution. Group 3 data were presented separately.
Time Frame: 30 days after the vaccination with MenACYW Conjugate or Menveo® vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS2. Here, "overall number of participants analyzed" = participants with available data for this outcome measure and 'Number analyzed'=participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Group 2: Menveo® Vaccine (Mexico): Participants aged 2 months (at the time of enrollment) received Menveo® vaccine at the age of Months 2, 4, 6, and 12 along with Prevnar 13®, Hexacima®, vaccines at the age of Months 2, 4, 6 and 12; RotaTeq® vaccine at the age of Months 2, 4 and 6 and and MMR®II vaccine at the age of Month 12.
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico)
Number analyzed (Participants) | 57 | 25
titers
  Serogroup A | 1102 [808 to 1502] | 5113 [2999 to 8717]
  Serogroup C | 2023 [1551 to 2639] | 572 [338 to 969]
  Serogroup Y | 1156 [913 to 1464] | 2288 [1343 to 3900]
  Serogroup W | 3135 [2196 to 4474] | 1938 [1075 to 3493]

40. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by rSBA Following Last Vaccination With MenACYW Conjugate Vaccine or Menveo® Vaccine: Group 3
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by rSBA. Titers were expressed in terms of 1/dilution.
Time Frame: 30 days after the vaccination with MenACYW Conjugate vaccine at the age of 12 months (i.e., at the age of 13 months)
Population: as for outcome 39
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 67
titers
  Serogroup A | 1234 [864 to 1762]
  Serogroup C | 236 [114 to 485]
  Serogroup Y | 586 [394 to 871]
  Serogroup W | 816 [464 to 1433]

41. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions After Any and Each Vaccination
Description: SR: expected AR (sign/symptom) observed & reported under conditions (nature & onset) prelisted (i.e., solicited) in protocol & CRF. Injection site reactions were tenderness, erythema & swelling. Assessment of injection site reactions after MenACYW Conjugate vaccine, Menveo, Prevnar 13, Hexacima, MMR, Pentaxim & ENGERIX-B allowed local reactogenicity assessment & helped to identify injection site reaction per vaccine received. Here, for Groups (Gps) 2 & 4: "0" in number analyzed for MenACYW vaccine (Vac.) categories signifies that no participant were evaluable; for Gps 1, 3 & 4: "0" in number analyzed for Menveo Vac. categories signifies that no participant were evaluable; for Gps 3 and 4: '0' in number analyzed field of Hexacima Vac. categories signifies that no participant were evaluable; for Gps 1 and 2: '0' in number analyzed field of Pentaxim and ENGERIX-B Vac. categories signifies that no participant were evaluable, as specified vaccines were not administered in specified groups.
Time Frame: Within 7 days after any vaccination and each vaccination (i.e., at the age 2 months, 3 months, 4 months, 4.5 months, 6 months and 12 months)
Population: Safety analysis set. 'Number analyzed'=participants with available data for each specified category & '0' in number analyzed field of specified age of vaccination (2, 3, 4, 4.5, 6 & 12 months) signifies that no participants received specified category vaccine & thus were not available for analysis. Reported AEs for each arm were presented as pre-specified in protocol & were not planned to be collected for Rotavirus vaccine because it was given orally & no injection site reactions were expected.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 201 | 99 | 150 | 75
Participants
  MenACYW conjugate vaccine: Tenderness: Post any vaccination: number analyzed (Participants) | 200 | 0 | 149 | 0
  MenACYW conjugate vaccine: Tenderness: Post any vaccination | 121 |  | 9 |
  MenACYW conjugate vaccine: Erythema: Post any vaccination: number analyzed (Participants) | 200 | 0 | 149 | 0
  MenACYW conjugate vaccine: Erythema: Post any vaccination | 52 |  | 11 |
  MenACYW conjugate vaccine: Swelling: Post any vaccination: number analyzed (Participants) | 200 | 0 | 149 | 0
  MenACYW conjugate vaccine: Swelling: Post any vaccination | 24 |  | 6 |
  Menveo: Tenderness: Post any vaccination: number analyzed (Participants) | 0 | 99 | 0 | 0
  Menveo: Tenderness: Post any vaccination |  | 60 |  |
  Menveo: Erythema: Post any vaccination: number analyzed (Participants) | 0 | 99 | 0 | 0
  Menveo: Erythema: Post any vaccination |  | 13 |  |
  Menveo: Swelling: Post any vaccination: number analyzed (Participants) | 0 | 99 | 0 | 0
  Menveo: Swelling: Post any vaccination |  | 9 |  |
  Prevnar 13: Tenderness: Post any vaccination: number analyzed (Participants) | 200 | 99 | 150 | 75
  Prevnar 13: Tenderness: Post any vaccination | 125 | 57 | 8 | 7
  Prevnar 13: Erythema: Post any vaccination: number analyzed (Participants) | 200 | 99 | 150 | 75
  Prevnar 13: Erythema: Post any vaccination | 48 | 20 | 9 | 4
  Prevnar 13: Swelling: Post any vaccination: number analyzed (Participants) | 200 | 99 | 150 | 75
  Prevnar 13: Swelling: Post any vaccination | 21 | 4 | 5 | 4
  Hexacima: Tenderness: Post any vaccination: number analyzed (Participants) | 200 | 99 | 0 | 0
  Hexacima: Tenderness: Post any vaccination | 132 | 56 |  |
  Hexacima: Erythema: Post any vaccination: number analyzed (Participants) | 200 | 99 | 0 | 0
  Hexacima: Erythema: Post any vaccination | 73 | 20 |  |
  Hexacima: Swelling: Post any vaccination: number analyzed (Participants) | 200 | 99 | 0 | 0
  Hexacima: Swelling: Post any vaccination | 32 | 7 |  |
  MMR: Tenderness: Post any vaccination: number analyzed (Participants) | 191 | 91 | 148 | 75
  MMR: Tenderness: Post any vaccination | 69 | 24 | 3 | 3
  MMR: Erythema: Post any vaccination: number analyzed (Participants) | 191 | 91 | 148 | 75
  MMR: Erythema: Post any vaccination | 66 | 27 | 5 | 3
  MMR: Swelling: Post any vaccination: number analyzed (Participants) | 191 | 91 | 148 | 75
  MMR: Swelling: Post any vaccination | 14 | 6 | 1 | 1
  Pentaxim: Tenderness: Post any vaccination: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Tenderness: Post any vaccination |  |  | 7 | 6
  Pentaxim: Erythema: Post any vaccination: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Erythema: Post any vaccination |  |  | 18 | 4
  Pentaxim: Swelling: Post any vaccination: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Swelling: Post any vaccination |  |  | 11 | 3
  ENGERIX-B: Tenderness: Post any vaccination: number analyzed (Participants) | 0 | 0 | 149 | 75
  ENGERIX-B: Tenderness: Post any vaccination |  |  | 5 | 3
  ENGERIX-B: Erythema: Post any vaccination: number analyzed (Participants) | 0 | 0 | 149 | 75
  ENGERIX-B: Erythema: Post any vaccination |  |  | 8 | 4
  ENGERIX-B: Swelling: Post any vaccination: number analyzed (Participants) | 0 | 0 | 149 | 75
  ENGERIX-B: Swelling: Post any vaccination |  |  | 5 | 1
  MenACYW conjugate vaccine: Tenderness: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 0 | 0 | 0
  MenACYW conjugate vaccine: Tenderness: Post vaccination at the age of 2 months | 87 |  |  |
  MenACYW conjugate vaccine: Erythema: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 0 | 0 | 0
  MenACYW conjugate vaccine: Erythema: Post vaccination at the age of 2 months | 19 |  |  |
  MenACYW conjugate vaccine: Swelling: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 0 | 0 | 0
  MenACYW conjugate vaccine: Swelling: Post vaccination at the age of 2 months | 9 |  |  |
  Menveo: Tenderness: Post vaccination at the age of 2 months: number analyzed (Participants) | 0 | 99 | 0 | 0
  Menveo: Tenderness: Post vaccination at the age of 2 months |  | 38 |  |
  Menveo: Erythema: Post vaccination at the age of 2 months: number analyzed (Participants) | 0 | 99 | 0 | 0
  Menveo: Erythema: Post vaccination at the age of 2 months |  | 6 |  |
  Menveo: Swelling: Post vaccination at the age of 2 months: number analyzed (Participants) | 0 | 99 | 0 | 0
  Menveo: Swelling: Post vaccination at the age of 2 months |  | 3 |  |
  Prevnar 13: Tenderness: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 150 | 75
  Prevnar 13: Tenderness: Post vaccination at the age of 2 months | 81 | 35 | 5 | 5
  Prevnar 13: Erythema: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 150 | 75
  Prevnar 13: Erythema: Post vaccination at the age of 2 months | 16 | 6 | 5 | 2
  Prevnar 13: Swelling: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 150 | 75
  Prevnar 13: Swelling: Post vaccination at the age of 2 months | 6 | 1 | 2 | 2
  Hexacima: Tenderness: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 0 | 0
  Hexacima: Tenderness: Post vaccination at the age of 2 months | 82 | 32 |  |
  Hexacima: Erythema: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 0 | 0
  Hexacima: Erythema: Post vaccination at the age of 2 months | 21 | 5 |  |
  Hexacima: Swelling: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 0 | 0
  Hexacima: Swelling: Post vaccination at the age of 2 months | 9 | 3 |  |
  MenACYW conjugate vaccine: Tenderness: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 0
  MenACYW conjugate vaccine: Tenderness: Post vaccination at the age of 3 months |  |  | 4 |
  MenACYW conjugate vaccine: Erythema: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 0
  MenACYW conjugate vaccine: Erythema: Post vaccination at the age of 3 months |  |  | 6 |
  MenACYW conjugate vaccine: Swelling: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 148 | 0
  MenACYW conjugate vaccine: Swelling: Post vaccination at the age of 3 months |  |  | 3 |
  Pentaxim: Tenderness: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Tenderness: Post vaccination at the age of 3 months |  |  | 3 | 2
  Pentaxim: Erythema: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Erythema: Post vaccination at the age of 3 months |  |  | 7 | 2
  Pentaxim: Swelling: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 148 | 75
  Pentaxim: Swelling: Post vaccination at the age of 3 months |  |  | 4 | 2
  Menveo: Tenderness: Post vaccination at the age of 4 months: number analyzed (Participants) | 0 | 94 | 0 | 0
  Menveo: Tenderness: Post vaccination at the age of 4 months |  | 36 |  |
  Menveo: Erythema: Post vaccination at the age of 4 months: number analyzed (Participants) | 0 | 94 | 0 | 0
  Menveo: Erythema: Post vaccination at the age of 4 months |  | 3 |  |
  Menveo: Swelling: Post vaccination at the age of 4 months: number analyzed (Participants) | 0 | 94 | 0 | 0
  Menveo: Swelling: Post vaccination at the age of 4 months |  | 3 |  |
  Prevnar 13: Tenderness: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Prevnar 13: Tenderness: Post vaccination at the age of 4 months | 71 | 32 |  |
  Prevnar 13: Erythema: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Prevnar 13: Erythema: Post vaccination at the age of 4 months | 21 | 4 |  |
  Prevnar 13: Swelling: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Prevnar 13: Swelling: Post vaccination at the age of 4 months | 8 | 2 |  |
  Hexacima: Tenderness: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Hexacima: Tenderness: Post vaccination at the age of 4 months | 77 | 33 |  |
  Hexacima: Erythema: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Hexacima: Erythema: Post vaccination at the age of 4 months | 26 | 4 |  |
  Hexacima: Swelling: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Hexacima: Swelling: Post vaccination at the age of 4 months | 15 | 2 |  |
  Prevnar 13: Tenderness: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Prevnar 13: Tenderness: Post vaccination at the age of 4.5 months |  |  | 5 | 4
  Prevnar 13: Erythema: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Prevnar 13: Erythema: Post vaccination at the age of 4.5 months |  |  | 5 | 2
  Prevnar 13: Swelling: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Prevnar 13: Swelling: Post vaccination at the age of 4.5 months |  |  | 3 | 2
  Pentaxim: Tenderness: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Tenderness: Post vaccination at the age of 4.5 months |  |  | 3 | 4
  Pentaxim: Erythema: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Erythema: Post vaccination at the age of 4.5 months |  |  | 7 | 2
  Pentaxim: Swelling: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Swelling: Post vaccination at the age of 4.5 months |  |  | 4 | 1
  MenACYW conjugate vaccine: Tenderness: Post vaccination at the age of 6 months: number analyzed (Participants) | 193 | 0 | 149 | 0
  MenACYW conjugate vaccine: Tenderness: Post vaccination at the age of 6 months | 75 |  | 6 |
  MenACYW conjugate vaccine: Erythema: Post vaccination at the age of 6 months: number analyzed (Participants) | 193 | 0 | 149 | 0
  MenACYW conjugate vaccine: Erythema: Post vaccination at the age of 6 months | 20 |  | 7 |
  MenACYW conjugate vaccine: Swelling: Post vaccination at the age of 6 months: number analyzed (Participants) | 193 | 0 | 149 | 0
  MenACYW conjugate vaccine: Swelling: Post vaccination at the age of 6 months | 7 |  | 2 |
  Menveo: Tenderness: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 93 | 0 | 0
  Menveo: Tenderness: Post vaccination at the age of 6 months |  | 31 |  |
  Menveo: Erythema: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 93 | 0 | 0
  Menveo: Erythema: Post vaccination at the age of 6 months |  | 4 |  |
  Menveo: Swelling: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 93 | 0 | 0
  Menveo: Swelling: Post vaccination at the age of 6 months |  | 1 |  |
  Prevnar 13: Tenderness: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 0 | 0
  Prevnar 13: Tenderness: Post vaccination at the age of 6 months | 75 | 30 |  |
  Prevnar 13: Erythema: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 0 | 0
  Prevnar 13: Erythema: Post vaccination at the age of 6 months | 21 | 10 |  |
  Prevnar 13: Swelling: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 0 | 0
  Prevnar 13: Swelling: Post vaccination at the age of 6 months | 8 | 1 |  |
  Hexacima: Tenderness: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 0 | 0
  Hexacima: Tenderness: Post vaccination at the age of 6 months | 73 | 30 |  |
  Hexacima: Erythema: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 0 | 0
  Hexacima: Erythema: Post vaccination at the age of 6 months | 32 | 11 |  |
  Hexacima: Swelling: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 0 | 0
  Hexacima: Swelling: Post vaccination at the age of 6 months | 11 | 2 |  |
  Pentaxim: Tenderness: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Tenderness: Post vaccination at the age of 6 months |  |  | 5 | 3
  Pentaxim: Erythema: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Erythema: Post vaccination at the age of 6 months |  |  | 11 | 3
  Pentaxim: Swelling: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Pentaxim: Swelling: Post vaccination at the age of 6 months |  |  | 5 | 2
  ENGERIX-B: Tenderness: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  ENGERIX-B: Tenderness: Post vaccination at the age of 6 months |  |  | 5 | 3
  ENGERIX-B: Erythema: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  ENGERIX-B: Erythema: Post vaccination at the age of 6 months |  |  | 8 | 4
  ENGERIX-B: Swelling: Post vaccination at the age of 6 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  ENGERIX-B: Swelling: Post vaccination at the age of 6 months |  |  | 5 | 1
  MenACYW conjugate vaccine: Tenderness: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 0 | 148 | 0
  MenACYW conjugate vaccine: Tenderness: Post vaccination at the age of 12 months | 77 |  | 4 |
  MenACYW conjugate vaccine: Erythema: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 0 | 148 | 0
  MenACYW conjugate vaccine: Erythema: Post vaccination at the age of 12 months | 27 |  | 3 |
  MenACYW conjugate vaccine: Swelling: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 0 | 148 | 0
  MenACYW conjugate vaccine: Swelling: Post vaccination at the age of 12 months | 11 |  | 2 |
  Menveo: Tenderness: Post vaccination at the age of 12 months: number analyzed (Participants) | 0 | 91 | 0 | 0
  Menveo: Tenderness: Post vaccination at the age of 12 months |  | 30 |  |
  Menveo: Erythema: Post vaccination at the age of 12 months: number analyzed (Participants) | 0 | 91 | 0 | 0
  Menveo: Erythema: Post vaccination at the age of 12 months |  | 9 |  |
  Menveo: Swelling: Post vaccination at the age of 12 months: number analyzed (Participants) | 0 | 91 | 0 | 0
  Menveo: Swelling: Post vaccination at the age of 12 months |  | 3 |  |
  Prevnar 13: Tenderness: Post vaccination at the age of 12 months: number analyzed (Participants) | 144 | 69 | 0 | 0
  Prevnar 13: Tenderness: Post vaccination at the age of 12 months | 50 | 21 |  |
  Prevnar 13: Erythema: Post vaccination at the age of 12 months: number analyzed (Participants) | 144 | 69 | 0 | 0
  Prevnar 13: Erythema: Post vaccination at the age of 12 months | 15 | 10 |  |
  Prevnar 13: Swelling: Post vaccination at the age of 12 months: number analyzed (Participants) | 144 | 69 | 0 | 0
  Prevnar 13: Swelling: Post vaccination at the age of 12 months | 10 | 2 |  |
  Hexacima: Tenderness: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 91 | 0 | 0
  Hexacima: Tenderness: Post vaccination at the age of 12 months | 79 | 29 |  |
  Hexacima: Erythema: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 91 | 0 | 0
  Hexacima: Erythema: Post vaccination at the age of 12 months | 37 | 16 |  |
  Hexacima: Swelling: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 91 | 0 | 0
  Hexacima: Swelling: Post vaccination at the age of 12 months | 16 | 2 |  |
  MMR: Tenderness: Post vaccination at the age of 12 months: number analyzed (Participants) | 191 | 91 | 148 | 75
  MMR: Tenderness: Post vaccination at the age of 12 months | 69 | 24 | 3 | 3
  MMR: Erythema: Post vaccination at the age of 12 months: number analyzed (Participants) | 191 | 91 | 148 | 75
  MMR: Erythema: Post vaccination at the age of 12 months | 66 | 27 | 5 | 3
  MMR: Swelling: Post vaccination at the age of 12 months: number analyzed (Participants) | 191 | 91 | 148 | 75
  MMR: Swelling: Post vaccination at the age of 12 months | 14 | 6 | 1 | 1

42. Secondary Outcome: Number of Participants With Solicited Systemic Reactions After Any and Each Vaccination
Description: A solicited reaction (SR) was an expected adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the case report form (CRF) and considered as related to the product administered. Solicited systemic reactions included fever, vomiting, crying abnormal, drowsiness, appetite lost, and irritability. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 7 days after any vaccination and each vaccination (i.e., at the age of 2 months, 3 months, 4 months, 4.5 months, 6 months and 12 months)
Population: Analysis was performed on safety analysis set. Here, 'Number analyzed'=participants with available data for each specified category and '0' in the number analyzed field signifies that none of the participants received the specified category vaccination and thus were not available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 201 | 99 | 150 | 75
Participants
  Fever: Post-any vaccination: number analyzed (Participants) | 199 | 98 | 149 | 75
  Fever: Post-any vaccination | 84 | 33 | 11 | 6
  Vomiting: Post-any vaccination: number analyzed (Participants) | 200 | 99 | 150 | 75
  Vomiting: Post-any vaccination | 39 | 11 | 6 | 0
  Crying abnormal: Post-any vaccination: number analyzed (Participants) | 200 | 99 | 150 | 75
  Crying abnormal: Post-any vaccination | 117 | 50 | 18 | 6
  Drowsiness: Post-any vaccination: number analyzed (Participants) | 200 | 99 | 150 | 75
  Drowsiness: Post-any vaccination | 80 | 36 | 33 | 17
  Appetite lost: Post-any vaccination: number analyzed (Participants) | 200 | 99 | 150 | 75
  Appetite lost: Post-any vaccination | 72 | 33 | 26 | 11
  Irritability: Post-any vaccination: number analyzed (Participants) | 200 | 99 | 150 | 75
  Irritability: Post-any vaccination | 134 | 58 | 32 | 20
  Fever: Post vaccination at the age of 2 months: number analyzed (Participants) | 198 | 97 | 149 | 75
  Fever: Post vaccination at the age of 2 months | 29 | 11 | 0 | 0
  Vomiting: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 150 | 75
  Vomiting: Post vaccination at the age of 2 months | 18 | 6 | 4 | 0
  Crying abnormal: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 150 | 75
  Crying abnormal: Post vaccination at the age of 2 months | 72 | 29 | 9 | 2
  Drowsiness: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 150 | 75
  Drowsiness: Post vaccination at the age of 2 months | 51 | 19 | 15 | 7
  Appetite lost: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 150 | 75
  Appetite lost: Post vaccination at the age of 2 months | 34 | 13 | 7 | 2
  Irritability: Post vaccination at the age of 2 months: number analyzed (Participants) | 200 | 99 | 150 | 75
  Irritability: Post vaccination at the age of 2 months | 92 | 44 | 13 | 6
  Fever: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Fever: Post vaccination at the age of 3 months |  |  | 0 | 1
  Vomiting: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Vomiting: Post vaccination at the age of 3 months |  |  | 0 | 0
  Crying abnormal: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Crying abnormal: Post vaccination at the age of 3 months |  |  | 6 | 0
  Drowsiness: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Drowsiness: Post vaccination at the age of 3 months |  |  | 9 | 4
  Appetite lost: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Appetite lost: Post vaccination at the age of 3 months |  |  | 5 | 1
  Irritability: Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Irritability: Post vaccination at the age of 3 months |  |  | 5 | 6
  Fever: Post vaccination at the age of 4 months: number analyzed (Participants) | 195 | 93 | 0 | 0
  Fever: Post vaccination at the age of 4 months | 28 | 17 |  |
  Vomiting: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Vomiting: Post vaccination at the age of 4 months | 12 | 5 |  |
  Crying abnormal: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Crying abnormal: Post vaccination at the age of 4 months | 61 | 30 |  |
  Drowsiness: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Drowsiness: Post vaccination at the age of 4 months | 36 | 21 |  |
  Appetite lost: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Appetite lost: Post vaccination at the age of 4 months | 30 | 12 |  |
  Irritability: Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 94 | 0 | 0
  Irritability: Post vaccination at the age of 4 months | 74 | 38 |  |
  Fever: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Fever: Post vaccination at the age of 4.5 months |  |  | 9 | 5
  Vomiting: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Vomiting: Post vaccination at the age of 4.5 months |  |  | 0 | 0
  Crying abnormal: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Crying abnormal: Post vaccination at the age of 4.5 months |  |  | 8 | 3
  Drowsiness: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Drowsiness: Post vaccination at the age of 4.5 months |  |  | 13 | 6
  Appetite lost: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Appetite lost: Post vaccination at the age of 4.5 months |  |  | 12 | 4
  Irritability: Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Irritability: Post vaccination at the age of 4.5 months |  |  | 17 | 10
  Fever: Post vaccination at the age of 6 months: number analyzed (Participants) | 190 | 92 | 149 | 75
  Fever: Post vaccination at the age of 6 months | 26 | 7 | 1 | 0
  Vomiting: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 149 | 75
  Vomiting: Post vaccination at the age of 6 months | 13 | 4 | 1 | 0
  Crying abnormal: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 149 | 75
  Crying abnormal: Post vaccination at the age of 6 months | 60 | 20 | 2 | 2
  Drowsiness: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 149 | 75
  Drowsiness: Post vaccination at the age of 6 months | 38 | 12 | 12 | 6
  Appetite lost: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 149 | 75
  Appetite lost: Post vaccination at the age of 6 months | 20 | 10 | 10 | 6
  Irritability: Post vaccination at the age of 6 months: number analyzed (Participants) | 194 | 93 | 149 | 75
  Irritability: Post vaccination at the age of 6 months | 77 | 26 | 10 | 10
  Fever: Post vaccination at the age of 12 months: number analyzed (Participants) | 191 | 91 | 148 | 75
  Fever: Post vaccination at the age of 12 months | 39 | 9 | 1 | 0
  Vomiting: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 91 | 148 | 75
  Vomiting: Post vaccination at the age of 12 months | 10 | 2 | 1 | 0
  Crying abnormal: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 91 | 148 | 75
  Crying abnormal: Post vaccination at the age of 12 months | 60 | 21 | 4 | 2
  Drowsiness: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 91 | 148 | 75
  Drowsiness: Post vaccination at the age of 12 months | 33 | 14 | 6 | 7
  Appetite lost: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 91 | 148 | 75
  Appetite lost: Post vaccination at the age of 12 months | 43 | 16 | 11 | 3
  Irritability: Post vaccination at the age of 12 months: number analyzed (Participants) | 192 | 91 | 148 | 75
  Irritability: Post vaccination at the age of 12 months | 75 | 26 | 13 | 3

43. Secondary Outcome: Number of Participants With Unsolicited Adverse Events After Any and Each Vaccination
Description: An AE was any untoward medical occurrence in a participant or in a clinical investigation participant administered a medicinal product and which did not had any casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 30 days after any vaccination and each vaccination (i.e., at the age 2 months, 3 months, 4 months, 4.5 months, 6 months and 12 months)
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 201 | 99 | 150 | 75
Participants
  Post-any vaccination | 100 | 47 | 15 | 6
  Post vaccination at the age of 2 months | 33 | 15 | 5 | 3
  Post vaccination at the age of 3 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Post vaccination at the age of 3 months |  |  | 4 | 1
  Post vaccination at the age of 4 months: number analyzed (Participants) | 196 | 95 | 0 | 0
  Post vaccination at the age of 4 months | 25 | 15 |  |
  Post vaccination at the age of 4.5 months: number analyzed (Participants) | 0 | 0 | 149 | 75
  Post vaccination at the age of 4.5 months |  |  | 5 | 0
  Post vaccination at the age of 6 months: number analyzed (Participants) | 195 | 94 | 149 | 75
  Post vaccination at the age of 6 months | 45 | 23 | 4 | 3
  Post vaccination at the age of 12 months: number analyzed (Participants) | 193 | 91 | 148 | 75
  Post vaccination at the age of 12 months | 43 | 17 | 5 | 1

44. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events of Special Interests (AESIs)
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI was an event for which ongoing monitoring and rapid communication by the Investigator to the Sponsor must be done. Such an event might warrant further investigation in order to characterize and understand it. Depending on the nature of the event, rapid communication by the study Sponsor to other parties (e.g, regulators) might also be warranted. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: From Day 0 (i.e., before first vaccination, at the age of 2 months) up to 30 days post last vaccination at the age of 12 months in each Group (i.e., up to the age of 13 months)
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
Number analyzed (Participants) | 201 | 99 | 150 | 75
Participants
  SAE | 4 | 3 | 4 | 2
  AESI | 1 | 1 | 1 | 0

45. Secondary Outcome: Percentage of Participants With hSBA Titers Distribution Less Than (<) 1:4, 1:4 and 1:8 Against Meningococcal Serogroups A, C, Y and W Following Last Vaccination With MenACYW Conjugate or Menveo® Vaccine: Groups 1, 2 and 3 (up to Infant Age of 6 Months)
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Percentage of participants with hSBA Titers distribution < 1:4, 1:4 and 1:8 is reported in this outcome measure. Infant series here denotes the vaccines administered at the age of 6 months of participants.
Time Frame: 30 days after the vaccination at the age of 6 months of the infant series (i.e., at the age of 7 months)
Population: Analysis was performed on PPAS1. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 176 | 81 | 97
percentage of participants
  Serogroup A: <1:4 | 4.0 | 14.8 | 6.2
  Serogroup A: 1:4 | 5.1 | 16.0 | 15.5
  Serogroup A: 1:8 | 4.5 | 11.1 | 8.2
  Serogroup C: <1:4 | 0 | 1.2 | 5.2
  Serogroup C: 1:4 | 0 | 1.2 | 0
  Serogroup C: 1:8 | 0 | 9.9 | 0
  Serogroup Y: <1:4 | 0.6 | 1.2 | 5.2
  Serogroup Y: 1:4 | 0 | 1.2 | 2.1
  Serogroup Y: 1:8 | 0 | 1.2 | 3.1
  Serogroup W: <1:4 | 0.6 | 0 | 5.2
  Serogroup W: 1:4 | 0 | 0 | 0
  Serogroup W: 1:8 | 0 | 1.2 | 1.0

46. Secondary Outcome: Percentage of Participants With hSBA Titers Distribution <1:4, 1:4 and 1:8 Against Meningococcal Serogroups A, C, Y, and W Following Last Vaccination With MenACYW Conjugate or Menveo® Vaccine: Groups 1, 2 and 3
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. Percentage of participants with hSBA Titers distribution < 1:4, 1:4 and 1:8 is reported in this outcome measure.
Time Frame: 30 days after the vaccination at the age of 12 months (i.e., at the age of 13 months)
Population: Analysis was performed on PPAS1. Here, 'Number analyzed'=participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation)
Number analyzed (Participants) | 126 | 60 | 96
percentage of participants
  Serogroup A: <1:4 | 1.6 | 3.3 | 2.1
  Serogroup A: 1:4 | 0.8 | 1.7 | 8.3
  Serogroup A: 1:8 | 0.8 | 10.0 | 15.6
  Serogroup C: <1:4 | 0 | 3.3 | 8.3
  Serogroup C: 1:4 | 0.8 | 3.3 | 9.4
  Serogroup C: 1:8 | 0 | 5.0 | 1.0
  Serogroup Y: <1:4: number analyzed (Participants) | 125 | 60 | 96
  Serogroup Y: <1:4 | 0 | 0 | 16.7
  Serogroup Y: 1:4: number analyzed (Participants) | 125 | 60 | 96
  Serogroup Y: 1:4 | 0 | 0 | 3.1
  Serogroup Y: 1:8: number analyzed (Participants) | 125 | 60 | 96
  Serogroup Y: 1:8 | 0 | 0 | 0
  Serogroup W: <1:4: number analyzed (Participants) | 125 | 60 | 96
  Serogroup W: <1:4 | 0 | 0 | 14.6
  Serogroup W: 1:4: number analyzed (Participants) | 125 | 60 | 96
  Serogroup W: 1:4 | 0 | 0 | 5.2
  Serogroup W: 1:8: number analyzed (Participants) | 125 | 60 | 96
  Serogroup W: 1:8 | 0 | 0 | 1.0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: from Day 0 (before first vaccination, at the age of 2 months) up to 30 days post any vaccination. SRs: within 7 days post any vaccination. SAE: from Day 0 (i.e., before first vaccination, at the age of 2 months) up to 30 days post last vaccination at the age of 12 months in each group (i.e., up to the age of 13 months)
Description: SR: defined as an "expected" AR (sign or symptom) observed and reported under conditions prelisted (i.e., solicited) in protocol and CRF and considered as related to vaccination. Unsolicited AE: an observed AE that did not fulfill conditions of solicited reactions prelisted in the CRF in terms of diagnosis and/or onset window post-vaccination. Safety population. In AE section, SR: fever, crying abnormal, and appetite lost are reported under pyrexia, crying, and decreased appetite, respectively.
Arm/Group | Group 1: MenACYW Conjugate Vaccine (Mexico) | Group 2: Menveo® Vaccine (Mexico) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) | Group 4: Routine Pediatric Vaccines (Russian Federation)
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/99 | 0/150 | 0/75
Serious Adverse Events (participants affected / at risk) | 4/201 | 3/99 | 4/150 | 2/75
Other Adverse Events (participants affected / at risk) | 181/201 | 78/99 | 64/150 | 34/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (Mexico) (N=201) | Group 2: Menveo® Vaccine (Mexico) (N=99) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) (N=150) | Group 4: Routine Pediatric Vaccines (Russian Federation) (N=75)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atonic Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine Cell Hyperplasia Of Infancy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (Mexico) (N=201) | Group 2: Menveo® Vaccine (Mexico) (N=99) | Group 3: MenACYW Conjugate Vaccine (Russian Federation) (N=150) | Group 4: Routine Pediatric Vaccines (Russian Federation) (N=75)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 6 (7) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 41 (55) | 14 (20) | 6 (6) | 0 (0) — Vomiting events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Crying (General disorders) | 117 (253) | 50 (100) | 18 (29) | 6 (9)
Injection Site Erythema (General disorders) | 106 (321) | 38 (115) | 26 (64) | 8 (18)
Injection Site Haematoma (General disorders) | 5 (5) | 5 (6) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 142 (896) | 62 (401) | 15 (43) | 10 (24)
Injection Site Swelling (General disorders) | 38 (124) | 16 (31) | 14 (31) | 4 (11)
Pyrexia (General disorders) | 85 (126) | 38 (56) | 12 (12) | 7 (7) — Pyrexia/Fever events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Influenza (Infections and infestations) | 14 (16) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 31 (43) | 19 (26) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 29 (31) | 10 (10) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 72 (127) | 33 (51) | 26 (45) | 11 (16)
Somnolence (Nervous system disorders) | 80 (158) | 36 (66) | 33 (55) | 17 (30)
Irritability (Psychiatric disorders) | 134 (318) | 58 (134) | 32 (58) | 20 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03630705/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT03630705/SAP_001.pdf